CLINICAL TRIAL: NCT06594328
Title: Evaluating the Effect of Text Message Interventions in Maintaining Gingival Health in Pregnant Women: a Pragmatic Trial
Brief Title: Effect of Text Message Interventions in Maintaining Gingival Health in Pregnant Women
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Saima Chaudhry, Director CHPL, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UCD/ERCA/24/525
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Oral Health; Pregnancy
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mHealth (Experimental): participants of intervention group will receive text message reminder once a week on their mobile phones to brush and floss properly for the study duration
  Interventions: Behavioral: mHealth
- Non mHealth (No Intervention): Participants of non-intervention group will not receive text message reminder once a week on their mobile phones to brush and floss properly for the study duration

INTERVENTIONS:
Behavioral: mHealth — participants of intervention group will receive text message reminder once a week on their mobile phones to brush and floss properly for the study duration
  Arms: mHealth

SUMMARY:
Gingivitis is a common condition, affecting more than 60% of pregnant women due to hormonal changes and inadequate plaque control. Left untreated, gingivitis can lead to more serious periodontal diseases and systemic inflammation, posing risks to overall health and reducing quality of life. Therefore, the study aims to assess the effectiveness of text messages in maintaining gingival health in pregnant women. The primary objective is to determine whether these reminders, which focus on proper brushing and flossing techniques, can reduce gingivitis and improve overall oral hygiene during pregnancy.

This research follows a two-group, parallel-arm, single-blind randomized control trial (RCT) design. The trial will be conducted at the Department of Gynecology and Obstetrics at the University of Lahore Teaching Hospital. Eligible participants are adult pregnant women showing signs of gingivitis, excluding those with bleeding disorders or moderate to severe pre-existing periodontal disease. Participants are randomly assigned to either a control group or an intervention group using computer-generated randomization.

Both groups will undergo oral health assessments at baseline, using the Plaque Index (PI), Gingival Index (GI), and Bleeding on Probing (BOP) measures to gauge plaque buildup and gingival inflammation. Follow-up assessments will be conducted at 4-6 weeks and 12-16 weeks. The intervention group will receive a weekly text message reminding them to practice proper oral hygiene, such as brushing and flossing. Both groups will also receive in-person demonstrations of oral hygiene techniques to ensure standardized knowledge on effective oral care.

ELIGIBILITY:
Inclusion Criteria:

* Adult pregnant female in 2nd trimester.
* Access to a personal mobile phone.
* Suffering from gingivitis (> 10% sites with bleeding on probing)

Exclusion Criteria:

* Bleeding disorders.
* Pre-existing moderate to severe periodontal disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Oral Health Status | 1 year
  Gingival index will be used to measure the oral health status of the mHealth and nonmHealth groups. The index is scored from 0-4. Once the scaling and root planning is done, half of the participants will be given mhealth message and half will not be given any message. After every three months the gingival index will be measured and compared to baseline (one achieved after treatment). The outcome is the maintenance of the gingival index at the same level post treatment or its improvement. Any deterioration will be considered a negative outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Saima Chaudhry, Study Chair — University of Lahore
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No